CLINICAL TRIAL: NCT07334574
Title: A Safety, Tolerability and Efficacy Study of XP-006 Personalized Tumor mRNA Vaccine for Relapsed or Refractory B-Cell Non-Hodgkin's Lymphoma
Brief Title: Clinical Study of XP-006 mRNA Vaccine for R/R B-NHL
Acronym: XP-006
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Shanghai Xinpu BioTechnology Company Limited (Unknown)
Responsible Party: Principal Investigator, Zhao Weili, Professor, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025PCV006-XP006
Record Dates: First submitted 2026-01-03; First posted 2026-01-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: B-cell Non-Hodgkin's Lymphoma (B-NHL)
Keywords: B-cell non-Hodgkin's lymphoma; XP-006; Personalized; Neoantigen
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoantigen tumor vaccine monotherapy arm (Experimental): Dose Escalation and Randomization Phase vaccine: 0.2mg, 0.4mg, 1 mg. Dose Expansion Phase vaccine: MTD or 1mg. 3 weeks as a treatment cycle, a total of 9 cycles.
  Interventions: Biological: Personalized neoantigen tumor vaccine

INTERVENTIONS:
Biological: Personalized neoantigen tumor vaccine — Neoantigen tumor vaccine
  Other Names: XP-006

SUMMARY:
The main objective of this study is to observe and evaluate the safety and tolerability of the XP-006 personalized tumor mRNA vaccine for the treatment of relapsed or refractory B-cell non-Hodgkin's lymphoma. Secondary objectives focus on evaluating preliminary efficacy through several parameters: XP-006-induced antigen-specific CD4+/CD8+ T cell activation levels, objective remission rate (ORR), complete remission rate (CRR), disease control rate (DCR), duration of response (DOR), progression-free survival (PFS), and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily signed written informed consent files, able to comply with the study protocol, in the investigator's judgment.
2. Subjects must be ≥18 years of age at time of informed consent, regardless of gender.
3. B-NHL was confirmed by histology according to world Health Organization (WHO) disease classification (excluding primary central lymphoma and HIV-associated lymphoma).
4. Prior treatment with sufficient first-line anti-lymphoma therapy, no remission within 90 days of the last administration, or disease progression after sufficient first-line anti-lymphoma therapy, and no current anti-lymphoma therapy (≥2 weeks since the last anti-lymphoma therapy). Patients were allowed to receive hormone drugs or rituximab at least 1 week after enrollment for symptom control reasons.
5. Gene mutation and the peripheral blood HLA typing both meet the requirements of the vaccine.
6. There are evaluable lesions detected by PET/CT.
7. Life expectancy of more than 3 months.
8. ECOG 0-2 points.
9. No serious organic lesions in the main organs, meeting the requirements of the following laboratory examination indicators (conducted within 7 days before treatment) : ① Absolute value of neutrophil count ≥1500/mm3; Platelet count ≥75,000/mm3 ② Total bilirubin ≤2× upper limit of normal value (ULN) ③ Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) (serum glutamate pyruvate aminotransferase [SGPT]) ≤3× upper limit of normal value (ULN) ④ the creatinine clearance rate was ≥60ml/min ⑤ No cardiac dysfunction.

Exclusion Criteria:

1. Pregnant or lactating women (lactating women must agree not to breastfeed while taking pomadomide);
2. Known hepatitis B (HBV), hepatitis C (HCV) infection (HBV infection refers to HBV-DNA > detectable limit); And other acquired, congenital immune deficiency disorders, including but not limited to HIV-infected persons;
3. Subjects with a history of deep vein thrombosis (DVT) or pulmonary embolism (PE) within the past 12 months;
4. Bone marrow failure, defined as ANC<1500/mm3 or platelet <75,000/mm3, unless hematologic changes are thought to be associated with lymphomas infiltrating the bone marrow;
5. Clinically significant heart disease, including unstable angina, acute myocardial infarction 6 months before enrollment, congestive heart failure (NYHA) heart function grade III or IV; Or left ventricular ejection fraction <50%;
6. Lymphoma with central nervous system (CNS) involvement;
7. Those who are known to be allergic to the test drug ingredients;
8. Those who have received grade II or above surgery within three weeks before treatment;
9. Patients who have received organ transplants;
10. Has been diagnosed with or is being treated for malignancy other than lymphoma, except for: ① They have received therapeutic treatment and have not had known active disease malignancy for ≥5 years prior to enrollment; ② Basal cell carcinoma of the skin (except melanoma) without signs of disease after adequate treatment; ③ Cervical carcinoma in situ without signs of disease after adequate treatment.
11. With severe infection;
12. Substance abuse, medical, psychological, or social conditions that may interfere with the subjects' participation in the study or evaluation of the study results; The researchers deemed unsuitable for the group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) & Maximum tolerated dose (MTD) | Day1 to Day 21

SECONDARY OUTCOMES:
Objective remission rate at the end of treatment | Up to approximately 2 years
Progression-Free Survival (PFS) | Up to approximately 2 years
  Progression-free Survival of Personalized mRNA Tumor Vaccine
Overall Survival (OS) | Up to approximately 2 years
  Overall Survival of Personalized mRNA Tumor Vaccine
Reaction of antigen-specific T cells in peripheral blood | Up to 104 weeks
  personalized tumor vaccine induced neoantigen-specific CD4+ and CD8+ T lymphocyte responses

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No